CLINICAL TRIAL: NCT04585529
Title: Flows of Emergency Surgery and Delay in Admission to the Operating Room: a Multicenter Prospective Observational Study in France
Brief Title: Surgical Emergency Flows and Delays in Admission to the Operating Room
Acronym: ACUTE-FLOW
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: NI2020/01
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Surgery; Emergencies; Postoperative Complications
Keywords: delay; organization
MeSH Terms: conditions — Emergencies; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
French hospitals treat non-elective surgery according to three organizational models: in a dedicated multi-specialty emergency operative room (OR), in a dedicated OR within a specialized surgical platform or in any available OR from a list of non-dedicated OR. Some triage algorithms for the classification of non-elective surgery have been described but are not routinely applied. The rate of delay in the management of non-elective surgery in France is not known. Reducing this delay decreased mortality and morbidity in urgent surgery (McIsaac D, et al., CMAJ 2017). Optimizing the flow of non-elective surgery represents a major challenge. The main objective of this study is to determine the rate of delay in admission to the OR in emergency surgery through a multicenter prospective observational study in France. All patients requiring urgent surgical management (<72 hours) will be included. The ideal time for surgery was previously defined by surgeons according to the NEST classification (NEST 1: within minutes; NEST 2: < 1 hour; NEST 3: < 4 hours; NEST 4: < 12 hours; NEST 5: < 48 hours; NEST 6: < 72 hours). For each patient, the ratio between the observed time (actual Time To Surgery [aTTS] ) and the ideal time (ideal Time To Surgery [iTTS]) will be determined. The delay is identified by aTTS/iTTS ratio >1.

ELIGIBILITY:
Inclusion Criteria:

any patient meeting the Following two criteria

* at least 18 ys old
* decision for unplanned surgery (which should be performed within 72 hours according to the protocol)
* in one of the following hospitals: Lille University hospital, Grenoble University hospital, Strasbourg University hospital, Paris University hospitals (Européen Georges Pompidou, Beaujon, H. Mondor), Lyon University hospital (Hôpital E. Herriot, Lyon Sud), Angers University hospital, Anthony Private hospital).

Exclusion Criteria:

* obstetrics
* interventional radiology
* endoscopies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged at least 18 years hospitalized and requiring non-elective surgery.
  Non-elective means that the surgery must ideally be performed within 72 hours. Patients may be coming in via the emergency department or may already be hospitalized when requiring surgical intervention.
  Anthony).
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of OR admission delay (delay = aTTS / iTTS > 1) | 30 days
  hours

SECONDARY OUTCOMES:
OR Admission delay according to the three organizational model | 30 days
  hours
OR Admission delay according to the period of work (day, night, and week-end) | 30 days
  hours
OR Admission delay according to the NEST classification | 30 days
  hours
delays related to organisational causes | 30 days
  hours
delays related to material causes | 30 days
  hours
delays related to human causes | 30 days
  hours
Impact of the delay on ICU length of stay | 30 days
  days
Impact of the delay on hospital length of stay | 30 days
  days
Impact of the delay on mortality | 30 days
Impact of the delay on morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Delphine GARRIGUE, MD, Principal Investigator — University Hospital, Lille, France; Benoit TAVERNIER, MD, PhD, Study Chair — University Hospital, Lille, France
Locations (10):
- France (10):
  - University hospital, Angers
  - Clinique, Antony
  - Beaujon Hospital, Clichy
  - Henri Mondor Hospital, Créteil
  - University Hospital, Grenoble
  - University hospital, Lille
  - Edouard Herriot Hospital, Lyon
  - Hôpital sud, Lyon
  - HEGP, Paris
  - University Hospital, Strasbourg